CLINICAL TRIAL: NCT05485753
Title: An Open, Multicenter, Phase Ib/II Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics/Pharmacodynamics, and Antitumor Activity of Tetra-specific Antibody GNC-038 Injection in Patients With Relapsed or Refractory Primary Central Nervous System Lymphoma (PCNSL) and Relapsed or Refractory Secondary Central Nervous System Lymphoma (SCNSL)
Brief Title: A Study of GNC-038, a Tetra-specific Antibody, in Patients With Central Nervous System Lymphoma (PCNSL) and Relapsed or Refractory Secondary Central Nervous System Lymphoma (SCNSL)
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sichuan Baili Pharmaceutical Co., Ltd. (Industry)
Collaborators: SystImmune Inc. (Industry); Baili-Bio (Chengdu) Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GNC-038-103
Record Dates: First submitted 2022-07-31; First posted 2022-08-03 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Primary Central Nervous System Lymphoma; Secondary Central Nervous System Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study treatment (Experimental): Participants receive GNC-038 as intravenous infusion for the first cycle (2 weeks). Participants with clinical benefit could receive additional treatment for more cycles. The administration will be terminated because of disease progression or intolerable toxicity occurring or other reasons.
  Interventions: Drug: GNC-038

INTERVENTIONS:
Drug: GNC-038 — Administration by intravenous infusion

SUMMARY:
In this study, the safety and preliminary efficacy of GNC-038 in patients with r relapsed or refractory primary central nervous system lymphoma (PCNSL) and relapsed or refractory secondary central nervous system lymphoma (SCNSL) will be investigated to assess the dose-limiting toxicity (DLT), maximum tolerated dose (MTD) or maximum administered dose (MAD) for MTD is not reached of GNC-038. The recommended dose for phase II (RP2D) clinical study will also be determined.

ELIGIBILITY:
Inclusion Criteria:

* 1. The subject can understand the informed consent, participate in and sign the informed consent voluntarily;
* 2. No gender limitation;
* 3. Age: ≥18;
* 4. Expected survival time ≥3 months;
* 5. Patients with primary CNS lymphoma (PCNSL) and secondary CNS lymphoma (SCNSL) confirmed by histology or cytology;
* 6. A. Patients with recurrent/refractory primary central nervous system lymphoma (PCNSL) and recurrent/refractory secondary central nervous system lymphoma (SCNSL) may be associated with ocular lymphoma;B. Patients with relapsed or refractory primary CNS lymphoma (PCNSL) and relapsed or refractory secondary CNS lymphoma (SCNSL) who were not eligible or intolerant to other therapies were determined by the investigator;Recurrence and refractory are defined as follows: Recurrence refers to the emergence of new lesions after adequate treatment to complete response (CR).Refractory refers to a patient who has experienced at least first-line treatment without disease remission, e.g. induction chemotherapy with methotrexate without CR.
* 7. KPS score ≥60;
* 8. Adverse reactions of previous antitumor therapy returned to CTCAE 5.0 grade ≤1 (except for the indicators that the researchers considered to be related to the disease, such as anemia, and toxicities that the researchers determined to be without safety risk, such as alopecia, grade 2 peripheral neurotoxicity, hypothyroidism stabilized by hormone replacement therapy, etc.);
* 9. Before the first administration, the organ function level should meet the following requirements:

Bone marrow function: In the absence of blood transfusion, G-CSF (long-acting white needle within 2 weeks) and medication correction within 7 days prior to screening:

Absolute neutrophil count (ANC) ≥15×10^9/L (subjects with bone marrow infiltration should be ≥0.5×10^9/L);Hemoglobin ≥90 g/L;Platelet count ≥90×10^9/L; Liver function: Total bilirubin ≤1.5 ULN (Gilbert's syndrome ≤3 ULN), transaminase (AST/ALT) ≤2.5 ULN (≤5.0 ULN for subjects with tumor invasive changes in the liver) without correction with hepatoprotective drugs within 7 days prior to screening; Renal function: Creatinine (Cr) ≤1.5 ULN and creatinine clearance (Ccr) ≥50 mL /min according to the Cockcroft and Gault formula; Routine urine / 24-hour urine protein quantification: qualitative urine protein ≤1+ (if qualitative urine protein ≥2+, 24-hour urine protein < 1g can be included); Cardiac function: left ventricular ejection fraction ≥50%; Coagulation function: fibrinogen ≥1.5g/L; Activated partial thrombin time (APTT) ≤1.5 ULN; Prothrombin time (PT) ≤1.5 ULN.

* 10. Fertile female subjects or male subjects with fertile partners must use highly effective contraception beginning 7 days before the first dose and up to 12 weeks after the last dose. Fertile female subjects must have a negative serum/urine pregnancy test within 7 days prior to initial dosing;
* 11. The subject is able and willing to follow the visits, treatment plans, laboratory tests, and other study-related procedures specified in the study protocol.

Exclusion Criteria:

* 1. Lung disease defined as grade ≥3 according to NCI-CTCAE V5.0; Patients with current interstitial lung disease (ILD) (except those who have recovered from previous interstitial pneumonia);
* 2. Active infections requiring systemic treatment, such as severe pneumonia, bacteremia, sepsis, etc.;
* 3. Active tuberculosis;
* 4. Brain stem tumor infiltration or only eye lesions;
* 5. Patients with active autoimmune diseases, such as: Systemic lupus erythematosus, systemic treatment of psoriasis, rheumatoid arthritis, inflammatory bowel disease, and hashimoto's thyroiditis, etc., with the exception of type I diabetes, only replacement therapy can control the hypothyroidism, no systemic treatment of skin disease (e.g., vitiligo, psoriasis), B cells caused by autoimmune disease;
* 6. Non-melanoma skin cancer in situ, superficial bladder cancer, cervical cancer in situ, gastrointestinal intramucosal cancer, breast cancer, localized prostate cancer and other cancers that have been cured and have not recurred within 5 years prior to the first administration are excluded;
* 7. HBsAg positive or HBcAb positive, and HBV-DNA test ≥ the upper limit of normal; HCV antibody positive and HCV-RNA≥ the upper limit of normal value; HIV antibody positive;
* 8. Poorly controlled hypertension (systolic blood pressure >150 mmHg or diastolic blood pressure >100 mmHg);
* 9. Have a history of serious cardiovascular and cerebrovascular diseases, including but not limited to: Severe cardiac rhythm or conduction abnormalities, such as ventricular arrhythmias and degree ⅲ ATrioventricular block requiring clinical intervention; Longer QT interval at rest (QTc > 450 msec for men or 470 msec for women); Acute coronary syndrome, congestive heart failure, aortic dissection, stroke, or other grade 3 or higher cardiovascular and cerebrovascular events occurred within 6 months prior to first administration; Heart failure with the New York Heart Association (NYHA) Heart function rating ≥II; 10. Patients with a history of allergy to recombinant humanized antibodies or to any excipient ingredient of GNC-038;
* 11. Pregnant or breastfeeding women;
* 12. Patients who cannot tolerate MRI examination;
* 13. Patients who underwent major surgery within 28 days prior to administration of the drug in this study, or who planned to undergo major surgery during the study period (except for puncture or biopsy surgery);
* 14. Prior organ transplantation or allogeneic hematopoietic stem cell transplantation (ALLO-HSCT);
* 15. Autologous hematopoietic stem cell transplantation (AUTO-HSCT) within 12 weeks prior to initiation of GNC-038 therapy;
* 16. Immunosuppressants are being used, including but not limited to: Cyclosporine, tacrolimus, etc. within 2 weeks prior to gnC-038 treatment; Gnc-038 received a high dose of glucocorticoid for 2 weeks prior to treatment (longer than 14 days, a steady dose of dexamethasone >5mg per day or equivalent dose of other glucocorticoids);
* 17. Received radiotherapy within 4 weeks prior to initiation of GNC-038 treatment;
* 18. Received anti-CD20 or anti-CD79B treatment within 4 weeks prior to initiation of GNC-038 and still responded;
* 19. Received chemotherapy and small molecule targeted therapy within 2 weeks prior to treatment;
* 20. Received CAR-T therapy within 12 weeks prior to initiation of GNC-038;
* 21. Participated in any other clinical trials within 4 weeks prior to administration of this trial;
* 22. Past or present central nervous system disease, including, but not limited to, stroke (imaging)
* 23. Medical examination indicated "lacunar cerebral infarction" except those requiring no treatment), severe brain injury, Senile dementia, Parkinson's disease, organic brain syndrome, psychosis;
* 24. Other conditions that the investigator considers inappropriate for participation in this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2023-02-10 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | Up to 17 days after the first dose
  The incidence and severity of adverse events during treatment were graded according to the National Cancer Institute Standard for Common Terminology for Adverse Events (NCI-CTCAE, v5.0).
Maximum tolerated dose (MTD) or maximum administrated dose (MAD) | Up to 17 days after the first dose
  In the dose increment stage, the highest dose whose estimated DLT rate is closest to the target DLT rate but does not exceed the upper bound of the equivalent interval of DLT rate is selected as MTD.
Treatment-Emergent Adverse Event (TEAE) | Up to approximately 36 months
  TEAE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally emerging, or any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition during the treatment of GNC-038. The type, frequency and severity of TEAE will be evaluated during the treatment of GNC-038.
The recommended dose for phase II clinical study（RP2D） | Up to 17 days after the first dose
  The RP2D is defined as the dose level chosen by the sponsor (in consultation with the investigators) for phase II study, based on safety, tolerability, efficacy, PK, and PD data collected during the dose escalation study of GNC-038.

SECONDARY OUTCOMES:
ORR (Objective Response Rate ) | Up to approximately 36 months
  ORR is defined as the percentage of participants, who has a CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions). The percentage of participants who experiences a confirmed CR or PR is according to RECIST 1.1.
PFS (Progression-free Survival) | Up to approximately 36 months
  The PFS is defined as the time from the participant's first dose of GNC-038 to the first date of either disease progression or death, whichever occurs first.
DCR (Disease Control Rate) | Up to approximately 36 months
  Number of patients showing Complete Response (CR, disappearance of all target lesions) or Partial Response (PR, at least a 30% decrease in the sum of longest diameter of target lesions taking as reference the baseline sum longest diameter) based on RECIST Criteria Version 1.0 (assessed by CT and/or MRI) for the best response.
DOR (Duration of Response) | Up to approximately 36 months
  The DOR for a responder is defined as the time from the participant's initial objective response to the first date of either disease progression or death, whichever occurs first.
CR (Complete Response) | Up to approximately 36 months
  Disappearance of all target lesions.
Adverse Events of special interest (AESI) | Up to approximately 36 months
  AESI is an event of scientific and medical interest specific to the sponsor's product or research project.
Peak Plasma Concentration（Cmax) | Up to 17 days after the first dose
  Maximum serum concentration (Cmax) of GNC-038 will be investigated.
Incidence and titer of ADA (Anti-drug antibody) | :Up to approximately 36 months
  Frequency and titer of anti-GNC-038 antibody (ADA) will be evaluated.
Incidence and titer of Nab | Up to approximately 36months
  Incidence and titer of Nab of GNC-038 will be evaluated.
Time to reach maximum concentration (Tmax) | Up to 17 days after the first dose
  Time to maximum serum concentration (Tmax) of GNC-038 will be investigated.
AUC0-inf | Up to 17 days after the first dose
  Area under the plasma concentration-time curve from time 0 extrapolated to infinite (AUC0-inf).
AUC0-t | Up to 14 days after the first dose of GNC-038
  Area under the plasma concentration-time curve from time 0 to last time of quantifiable concentration (AUC0-t).
Plasma clearance （CL） | Up to 17 days after the first dose
  To study the serum clearance rate of GNC-038 per unit time.
Elimination half life （T1/2） | Up to 17 days after the first dose
  Blood concentration - Area under time line.

CONTACTS AND LOCATIONS:
Overall Officials: Wenbin Li, Principal Investigator — Beijing Tiantan Hospital
Locations (4):
- China (4):
  - Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing GoBroad Boren Hospital, Beijing, Beijing Municipality
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan

IPD SHARING:
Plan to Share IPD: No